CLINICAL TRIAL: NCT07125508
Title: Tranexamic Acid for The Management of Bleeding Gastrointestinal Angioectasias: A Randomized, Placebo Controlled Trial
Brief Title: Tranexamic Acid for The Management of Bleeding Gastrointestinal Angioectasias
Acronym: TAMBA
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB # 4587
Record Dates: First submitted 2025-07-31; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Anemia; Small Bowel Bleeding; Angioectasias
Keywords: tranexamic acid; angioectasia
MeSH Terms: conditions — Anemia | interventions — Tranexamic Acid; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tranexamic Acid (Active Comparator): Patients randomized to the interventional arm will take oral tranexamic acid 650 mg three times per day for 3 months. They will have blood work drawn every month for the 3 month trial period.
  Interventions: Drug: Tranexamic Acid (TXA) treatment
- Placebo (Placebo Comparator): Patients randomized to the placebo comparator arm will take oral placebo medication three times per day for 3 months. They will have blood work drawn every month for the 3 month trial period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic Acid (TXA) treatment — Patients randomized to the interventional arm will take oral tranexamic acid 650 mg three times per day for 3 months. They will have blood work drawn every month for the 3 month trial period.
  Other Names: TXA
  Arms: Tranexamic Acid
Drug: Placebo — Placebo intervention
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if oral tranexamic acid works to treat gastrointestinal angioectasias. It will also learn about the safety of tranexamic acid. The main questions it aims to answer are:

Does tranexamic improve hemoglobin concentration and/or requirement for blood transfusions

What medical problems do participants have when taking tranexamic acid?

Researchers will compare tranexamic acid to a placebo (a look-alike substance that contains no drug) to see if it works to treat angioectasias.

Participants will:

Take tranexamic acid or a placebo three times per day, every day for 3 months Visit the clinic once per month for checkups and tests

DETAILED DESCRIPTION:
Currently, the mainstay of treatment for intestinal angioectasias (AEs) includes endoscopic ablation combined with octreotide and iron supplementation. However, many patients continue to suffer from persistent or recurrent symptomatic anemia and often require repeated hospitalizations for blood transfusions. Tranexamic acid (TXA) is a hemostatic agent that has the potential to be beneficial in patients with small bowel gastrointestinal bleeding. Through a literature review multiple case reports have highlighted the impact TXA treatment can have on patients with intestinal AEs. This study would help determine the potential additive effect of TXA in patients with symptomatic anemia due to gastrointestinal AEs. Further, the researchers seek to expand the applications of TXA with the goal of decreasing morbidity and mortality.

In the randomized control trial portion of the study, the researchers will enroll approximately 50 patients with diagnosed intestinal AEs through video capsule endoscopy and/or endoscopy who experience symptomatic anemia despite standard therapy including endoscopic ablation and iron supplementation. Subjects will be randomized to either the TXA treatment group versus the placebo treatment group for 3 months. Patients will have initial complete blood counts (CBC) measured as a baseline then subsequent CBCs measured at 1, 2 and 3 months. Patients will be monitored for drug side effects, symptoms related to anemia, the need for blood transfusions and hospitalizations related to gastrointestinal bleeding/anemia.

ELIGIBILITY:
Inclusion Criteria:

* Male, female, non-gender conforming patients aged >18 years with symptomatic anemia attributed to chronic gastrointestinal blood loss from angioectasias despite endoscopic ablation and iron therapy
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Contraindications to tranexamic acid (TXA) therapy
* Allergy to TXA, intracranial bleed, history of venous or arterial thromboembolism, active thromboembolic disease, ischemic retinopathy
* Bleeding/Coagulopathy disorder and/or on anticoagulation regimen
* Ulcerative colitis or Crohn's disease
* End stage renal disease
* Decompensated cirrhosis
* Pregnancy or intention to become pregnant
* Patient refusal of blood products because the secondary outcome is pre-determined
* Unable to give formal consent
* Participation in another interventional study where primary outcome includes hemoglobin/hematocrit values
* Inability to adhere to treatment regimen for 3 months
* Non-English speaking
* Patients < 18 years old

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-12-15 (Actual)

PRIMARY OUTCOMES:
Number of participants with improved hemoglobin concentrations and/or blood transfusions requirement | From enrollment to the end of treatment at 3 months
  To determine whether oral therapy with tranexamic results in improvement in serum hemoglobin concentration and/or requirement for blood transfusion compared to placebo in patients treated with standard endoscopic ablation and iron supplementation

SECONDARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events | From enrollment to the end of treatment at 3 months
  To determine the rate of clinically significant side effects associated with TXA therapy leading to drug withdrawal

CONTACTS AND LOCATIONS:
Locations (1):
- LSU Health Sciences Center - New Orleans, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-03): https://cdn.clinicaltrials.gov/large-docs/08/NCT07125508/Prot_SAP_000.pdf